CLINICAL TRIAL: NCT07016724
Title: Neoadjuvant Radiochemotherapy Combined With Cadonilizumab for Local Advanced Esophageal Squamous Cell Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Xiangbo Wan, Vice-president of the First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA2024-404-ESCC
Record Dates: First submitted 2025-02-11; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: cadonilizumab combined with neoadjuvant radiochemotherapy (Experimental): Subjects randomized in Arm 1 will be treated with cadonilizumab plus neoadjuvant radiochemotherapy before surgery.
  Interventions: Combination Product: cadonilizumab combined with neoadjuvant radiochemotherapy
- Arm 2: neoadjuvant radiochemotherapy (Placebo Comparator): Subjects randomized in Arm 2 will be treated with neoadjuvant radiochemotherapy before surgery.
  Interventions: Combination Product: neoadjuvant radiochemotherapy

INTERVENTIONS:
Combination Product: cadonilizumab combined with neoadjuvant radiochemotherapy — Subjects randomized to experimental arm will be treated with PD-1/CTLA-4 bi-antibody, termed as cadonilizumab, combined with neoadjuvant radiochemotherapy before surgery.
  Other Names: neoadjuvant radiochemotherapy
  Arms: Arm 1: cadonilizumab combined with neoadjuvant radiochemotherapy
Combination Product: neoadjuvant radiochemotherapy — Subjects in the arm 2, the control arm, will be treated with neoadjuvant radiochemotherapy.
  Arms: Arm 2: neoadjuvant radiochemotherapy

SUMMARY:
Esophageal squamous cell cancer (ESCC) has a high incidence in China. Although the fast development of immune check point inhibitors (ICIs), the rate of pCR is limited with the mode of ICIs combined with neoadjuvant radiochemotherapy. The rate of pCR under ICIs combined with neoadjuvant radiochemotherapy was reported around 50%, which means more than half of those patients could not obtain pCR in reality. In order to explore a more effective mode of neoadjuvant therapy for ESCC, we designed this study to evaluate the effect of PD-1/CTLA-4 bi-antibody, termed as cadonilizumab, combined with neoadjuvant radiochemotherapy in local advanced ESCC.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with esophageal squamous cell cancer;
* staged with cT1N+M0/cT2-3N0-3M0;
* experienced no cancer-related treatment;
* ECOG 0-1;
* Expected survival more than 6 months;
* aimed at neoadjuvant therapy for surger;
* have adquate organ function.

Exclusion Criteria:

* diagnosed with other types of cancer during last five years;
* have a tendency to bleed;
* accepted any type of cancer-related therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
pCR | perioperative
  pathological complete response

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbo Wan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- the First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No